CLINICAL TRIAL: NCT00169741
Title: Alterations in Renal Blood Flow as a Consequence of Percutaneous Nephrolithotomy (PERC)
Brief Title: Renogram Study With Percutaneous Nephrolithotomy (PERC): Alterations in Renal Blood Flow as a Consequence of PERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-043
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Renal Calculi
Keywords: Nephrolithiasis; Renal Calculi
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cohort (Other)
  Interventions: Other: Renogram

INTERVENTIONS:
Other: Renogram — Subjects who enroll in this study will undergo a nuclear scan called a renogram to assess renal function prior to surgery (baseline), approximately one hour after surgery (to assess percutaneous effects on renal function) and finally approximately 6 weeks post-operatively (to assess return to baseline).

SUMMARY:
Patients with large or otherwise complex renal calculi are commonly treated by percutaneous nephrolithotomy (PNL; PERC). PERC requires the creation of an approximately 10 mm channel through the renal parenchyma, into the intra-renal collecting system, in order to effect stone fragmentation and extraction. Although the nephrostomy tract is confined to a small fraction of the renal parenchyma (approximately 1%), the trauma associated with the creation of the tract will affect blood flow and oxygen delivery to regions beyond the immediate site of injury. It is possible that this could result in a significant functional renal impairment. There are several reports describing the effect of PERC on renal function, but interpretation of these studies is difficult, due to a lack of uniformity in patient selection and variability in the timing of peri-operative evaluation. Recent data from the investigators' lab, obtained from a porcine model, suggest that, acutely, PERC causes a significant decrease in renal function as measured by para amino hippurate (PAH) clearance. The purpose of this study is to determine, in a rigorous and standardized fashion, the acute effects of PERC on renal function, as measured by nuclear renography.

DETAILED DESCRIPTION:
PERC is a commonly used technique to treat patients harboring large or complex renal calculi. PERC is a particularly effective procedure, and has been associated with few complications. However, the effect PERC has on renal functional parameters is not well defined.

The effect of PERC on renal function has been examined in an animal model by several groups. In one porcine model, the baseline renal function, as defined by PAH and creatinine clearance, was compared to that measured at one month post-procedure. No acute data were recorded, but the authors did note that although there was no significant change in renal function at the one month follow-up point, there was a significant amount of renal scarring present. This finding of significant renal scarring following PERC in an animal model has been corroborated by others. One group has studied a canine model, and detected a significant diminution of renal function (defined by creatinine clearance) at 48 hours following PERC, and at 6 weeks following PERC renal function returned to normal. In human subjects undergoing PERC, percutaneous tracts have also been associated with renal scarring. These studies, both retrospective case series, did not capture strictly defined measures of renal function, such as creatinine clearance, but rather compared pre- and post-procedure serum creatinine as a surrogate for renal function. No significant change in serum creatinine was identified in either study, but blood collections were performed at variable times, in uncontrolled settings.

Nuclear renography is an imaging technique that records renal functional parameters. There has been only one report of nuclear renographic assessment of the effect of PERC on renal function. This report was an uncontrolled study, and the renograms were performed at a median of 22 days post-procedure. At this time interval, it is not possible to derive any conclusions regarding the acute effects of PERC on renal function.

The investigators have recently demonstrated in a porcine model that PERC is associated acutely with significant deleterious effects on renal function. Following routine PERC, glomerular filtration rate (GFR) and renal plasma flow (RPF) decline by 50% in both the treated and the untreated kidney and return to normal when measured at 72 & 74 hours (n=3 pigs). Sodium excretion, however, was markedly below baseline at 72 and 74 hours in 2 of the 3 pigs. PAH extraction, a measure of the efficiency of renal tubular secretion of organic anions, averaged 43.5 ± 9.7% and 42.6 ± 14.1% at 72 and 74 hours for the 3 pigs. These values are substantially below the baseline value of 80.4 ± 4.0% measured in sham-PNL pigs.

To date, the examination of the effect of PERC on renal function has been restricted to gross measures of function as defined by serum creatinine, and radionuclide studies performed at a sub-acute interval following PNL, often without differential measurements or controls. Importantly, the investigators' recent studies in a porcine model demonstrate that PERC may cause significant alterations in renal function. There is a need to define in a rigorous fashion the effect PERC has on renal blood flow and renal function. If a deleterious effect is identified, future efforts can be focused on minimizing this insult.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Methodist Urology in Indianapolis, IN
* Age greater than 18 years
* Ability to provide informed consent
* Unilateral renal calculi appropriate for percutaneous removal

Exclusion Criteria:

* Age less than 18
* Inability to give informed consent
* Pregnant
* Renal calculi associated with infection
* Serum creatinine > 1.4 mg/dL
* Renal obstruction
* Renal anatomic abnormality precluding accurate functional assessment using nuclear medicine techniques
* Renal duplication/anatomic abnormality (e.g., horseshoe kidney, malrotation, ectopia, etc.)
* Pre-existing diuretic therapy
* Solitary functional kidney or suspected significant differential in renal function
* Presence of diabetes, hypertension, or any other systemic disorder or medication known to affect renal function
* History of urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The hypothesis is that the effects of PERC anticipated on renal function will be largely resolved and the 6 week post-procedure study will not be significantly different from the pre-operative study. | One year after study completion

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States